CLINICAL TRIAL: NCT02657278
Title: The Influence of Peripheral Arterial Disease (PAD) on the Onset of Lactate Threshold (LT) in Patients Undergoing Cardiopulmonary Exercise Test (CPET)
Brief Title: Cardiopulmonary Exercise Test in Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Francesco Torella, Consultant Vascular Surgeon, Liverpool University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 825/15
Record Dates: First submitted 2016-01-13; First posted 2016-01-15 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral arterial disease,; Cardipulmonary Exercise Test
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Endovascular Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Symptomatic Peripheral arterial disease (Other): Patients scheduled to undergo surgery or angioplasty of the iliofemoral segment for intermittent claudication.
  Interventions: Procedure: Arterial Revascularization surgery or Endovascular procedure

INTERVENTIONS:
Procedure: Arterial Revascularization surgery or Endovascular procedure — Symptoms limited Cardiopulmonary Exercise Test (CPET) performed before and four weeks after surgical or endovascular correction of peripheral arterial disease

SUMMARY:
Aim: To determine whether the lactate threshold during CPET is influenced by the presence of haemodynamically significant PAD.

Assumption: Correction of haemodynamically significant PAD results in an increased LT, measured by CPET.

Design: Prospective study Population: Thirty patients scheduled to undergo surgical or percutaneous treatment of iliofemoral arterial disease for intermittent claudication.

DETAILED DESCRIPTION:
Patients scheduled to undergo surgery or angioplasty of the iliofemoral segment for intermittent claudication will be screened for inclusion. Consenting patients will undergo ABI measurements and CPET before treatment and four weeks after treatment. Study measures will be performed in the respiratory physiology laboratory at University Hospital Aintree. Demographic and medical details will be recorded including gender, age, smoking history and pack years, medical history and treatment and BMI. A record will be made of patuients' latest full blood count which will be routinely available in all participants before the procedure. Ankle-brachial index will be recorded. The subjects will undergo full CPET. This includes recording of baseline spirometry, full ECG monitoring throughout the test, measurement of ventilator parameters and recording of Borg breathlessness and leg fatigue score every minute. At the end of the test the reason for cessation will be documented. The test will be incremental with a 10-20W ramp determined according to baseline MVV aiming for the subject to exercise for 10-12 minutes. The test will involve 3 minutes rest, 2 minutes free-pedal followed by continuous ramping until volition. Recording will continue for 5 minutes recovery

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, ability to perform a CPET on a cycle ergometer, intermittent claudication as presenting complaint, age ≥18, iliofemoral arterial disease

Exclusion Criteria:

* Critical limb ischaemia, unwillingness to consent, previous amputation or other inability to perform CPET on a cycle ergometer, age <18, absence of iliofemoral arterial disease, any standard CPET exclusion based on American Thoracic Society/European Respiratory Society Guidelines, including severe arthritis or lower limb abnormality precluding exercise testing, severe hypertension at rest, unstable angina or acute coronary syndrome within the previous 6 weeks, terminal illness/advanced cancer or major psychiatric illness, including dementia, which precludes consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The difference in Lactate Threshold (LT) between the two CPETs | Four weeks following the intervention

SECONDARY OUTCOMES:
The correlation between rise in LT post treatment (if any) and haemodynamic measures of PAD improvement (ankle-brachial index - ABI - differential). | Four weeks following the intervention
The effect of the intervention on peak oxygen delivery during exercise. | Four weeks following the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Torella, Principal Investigator — Aintree University Hospital Foundation Trust
Locations (1):
- Liverpool Vascular & Endovascular Service and Department of Respiratory Medicine, Aintree University Hospitals NHS Foundation Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young EL, Karthikesalingam A, Huddart S, Pearse RM, Hinchliffe RJ, Loftus IM, Thompson MM, Holt PJ. A systematic review of the role of cardiopulmonary exercise testing in vascular surgery. Eur J Vasc Endovasc Surg. 2012 Jul;44(1):64-71. doi: 10.1016/j.ejvs.2012.03.022. Epub 2012 Apr 21. PMID 22521839
- [Derived] Barkat M, Key A, Ali T, Walker P, Duffy N, Snellgrove J, Torella F. Effect of treatment of peripheral arterial disease on the onset of anaerobic exercise during cardiopulmonary exercise testing. Physiol Rep. 2021 Apr;9(7):e14815. doi: 10.14814/phy2.14815. PMID 33818006
- [Derived] Key A, Ali T, Walker P, Duffy N, Barkat M, Snellgrove J, Torella F. Effect of peripheral arterial disease on the onset of lactate threshold during cardiopulmonary exercise test: study protocol. BMJ Open. 2016 Dec 19;6(12):e012763. doi: 10.1136/bmjopen-2016-012763. PMID 27993904